CLINICAL TRIAL: NCT06994832
Title: Examining Genetic Literacy and Numeracy in the General Population
Brief Title: Using Visual Arrays to Support Understanding of Genetic Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stephanie B. Seminara, MD (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Boston College (Other)
Responsible Party: Sponsor-Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, MGH Harvard Center for Reproductive Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2025P000889; P50HD104224 (NIH); NCT06905990 (obsolete NCT alias)
Record Dates: First submitted 2025-04-22; First posted 2025-05-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Decision Aid
Keywords: Lynch syndrome; colorectal cancer; colon cancer; genetic testing
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: One-to-one randomization into two parallel groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual Array (Experimental): Single, side-by-side visual array
  Interventions: Behavioral: Visual Array
- Narrative Visual Array (Experimental): Evolving narrative showing sequential visual arrays
  Interventions: Behavioral: Narrative Visual Array

INTERVENTIONS:
Behavioral: Visual Array — Single side-by-side visual array
  Arms: Visual Array
Behavioral: Narrative Visual Array — Evolving narrative with sequential visual arrays
  Arms: Narrative Visual Array

SUMMARY:
The goal of this study is to understand how people understand risk from genetic testing. The investigators want to understand what visual aid best helps people accurately assess risk. The investigators also want to understand how people relate risk to their health. The main questions the study aims to answer are:

1. Which visual aid most accurately show genetic risk?
2. How do people perceive risk related to genetic test results?
3. What factors are associated with people discussing their results with family?

Participants will:

1. receive of of two visual aids showing risk
2. state their estimation of risk
3. answer questions about how they feel about risk and sharing information with family

DETAILED DESCRIPTION:
This study aims to determine what visual aid helps people most accurately interpret risk from genetic test results. The study also examines how people perceive risk using the Tripartite Risk Model. Last, the study examines factors that are associated with intention to share genetic test results with family members.

Participants will provide brief sociodemographic information, complete brief health literacy and numeracy assessments, and questions about how they perceive risk. Participants will be informed of a genetic testing scenario and will receive one of two visual aids. After reviewing the visual aid, participants will state the risk shown in the visual aid and will answer questions about their perceived risk and sharing results with family members (blood relatives).

ELIGIBILITY:
Inclusion Criteria:

* ability to read and understand English
* opt-in consent

Exclusion Criteria:

* incorrect responses to validation questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1045 (Actual)
Dates: Start 2025-07-28 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Risk Accuracy | immediately after the intervention
  closest approximation to risk percentage depicted in the visual array

SECONDARY OUTCOMES:
Risk Perceptions | baseline
  Perceptions of deliberative, affective, and experiential risk using 7-point Likert-type scales
Communication Intent | immediately after the intervention
  Intent to communicate risk to blood relatives using 7-point Likert-type scale

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Dwyer, PhD, Principal Investigator — Boston College
Locations (1):
- Boston College, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared via the HarvardDataverse platform.
Time Frame: Start date: within one month of the publication of study results. End date: one year after posting.
Access Criteria: HarvardDataverse platform
URL: https://dataverse.harvard.edu/